CLINICAL TRIAL: NCT04617093
Title: A Post-Market Study of Performance and Safety of Low-flow Extracorporeal Carbon Dioxide Removal Using PrismaLung+ in Patients With Mild to Moderate Acute Respiratory Distress Syndrome
Brief Title: Post-Market Study of Low-flow ECCO2R Using PrismaLung+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXU542357
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mild to Moderate Acute Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Patient Population (Experimental): The planned PrismaLung+ treatment period for this study is 24 hours. Neuromuscular blockade and sedation will be required for the first 24 hours of ECCO2R treatment and thereafter, will be used at the discretion of the attending physician. Patients will require systemic anticoagulation with heparin during ECCO2R treatment. Blood warming during ECCO2R treatment will occur using the TherMax blood warmer.
  Interventions: Device: PrismaLung+

INTERVENTIONS:
Device: PrismaLung+ — Overall, up to 60 adult patients will be initiated on ECCO2R using PrismaLung+. A minimum of approximately 15 patients will be treated with ECCO2R using PrismaLung+ as standalone therapy and another minimum of approximately 15 patients will receive ECCO2R using PrismaLung+ in combination with CRRT.

SUMMARY:
PrismaLung+ is intended to provide extracorporeal carbon dioxide removal (ECCO2R) as a standalone therapy or in combination with continuous renal replacement therapy (CRRT). This study is a multi-centre, prospective, open-label, single-arm study. Adult patients with mild or moderate acute respiratory distress syndrome (ARDS) requiring mechanical ventilation were planned to receive ultra-lung protective ventilation (ULPV) associated with ECCO2R using PrismaLung+. The study will assess the capability of PrismaLung+ to allow ULPV, defined as a tidal volume (VT) of 4 mL/kg of predicted body weight, and confirm the safety of PrismaLung+.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is ≥ 18 years old
2. Patient is expected to receive ECCO2R for a minimum of 24 hours
3. Patient has mild or moderate ARDS according to the Berlin definition:

   * 100 mm Hg < PaO2/FiO2 ≤ 300 mm Hg, with PEEP ≥ 5 cm H2O, and
   * Bilateral lung opacities not fully explained by effusions, lobar/lung collapse, or nodules, and
   * Respiratory failure not fully explained by cardiac failure or fluid overload
4. Written informed consent to participate in the study from the patient, if possible, or from the identified authorized representative if the patient is unable to provide consent.

Exclusion Criteria:

1. Patients body weight < 30 kg
2. Patients with a contraindication for systemic anticoagulation with heparin
3. Patients with a platelet count < 50,000/µL
4. Patients on MV > 7 days
5. Patients with very severe, or stage 4 (as per GOLD staging System) chronic obstructive pulmonary disease (COPD)
6. Current or history of heparin-induced thrombocytopenia
7. Patients who are pregnant and/or breastfeeding
8. Patients not expected to survive the duration of the planned study treatment period (24 hours)
9. Patients currently participating in another interventional clinical study, except if the patient is in an investigational medicinal product study, already in follow-up without further administration of study drug, and has not received any investigational medicinal product within 5 half-lives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving ultra-lung protective ventilation (ULPV) 8 and 24 hours following ECCO2R initiation | 8 and 24 hours following ECCO2R initiation
  Must maintain PaCO2 < 50 mmHg. ULPV is defined as defined as a tidal volume (VT) of 4 mL/kg of predicted body weight.
Adverse Events related to study device | Day 1 to Day 28
  Adverse event related to the use of a study device. This definition includes AEs resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the study device.
  This definition includes any event resulting from use error or from intentional misuse of the study device.
Adverse Events related to study procedure | Day 1 to Day 28
  Adverse events related to the study procedure (ECCO2R or ECCO2R in combination with CRRT), irrespective of relatedness to the device.
Adverse Device Effect (ADE) | Day 1 to Day 28
  This includes study device and study procedure related adverse events.
Adverse Events leading to study withdrawal | Day 1 to Day 28
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in patients, users or other persons, in the context of a clinical investigation leading to study withdrawal.
Adverse events of special interest (AESIs) | Day 1 to Day 28
  The AESI's for this study include significant bleeding events (i.e. require administration of ≥ 1 unit of packed red blood cells (pRBC) or result in a related SAE).

SECONDARY OUTCOMES:
Carbon dioxide clearance after ECCO2R treatment | 8 hours following ECCO2R initiation
  CO2 clearance (mL/min) will be summarized descriptively by group and in total

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Investigational Site, Besançon
  - Investigational Site, Colombes
  - Investigational Site, Créteil
  - Investigational Site, Lille
  - Investigational Site, Marseille
  - Investigational Site, Montpellier
  - Investigational Site, Paris
  - Investigational Site, Strasbourg
  - Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Combes A, Levy B, Tapponnier R, Capellier G, Mekontso Dessap A, Duburcq T, Castelain V, Forel JM, Uhel F, Mayaux J, Goldstein J, Kurz J, Harenski K, Montgomery W, Parreno R, Jaber S. A prospective clinical evaluation of new ECCO2R technology in mild to moderate ARDS patients: assessing ultra-lung-protective ventilation with PRISMALUNG. Crit Care. 2026 Jan 6;30(1):15. doi: 10.1186/s13054-025-05827-4. PMID 41495763